CLINICAL TRIAL: NCT00118313
Title: Evaluation of Different Adjuvants for the Transdermal Administration of a Peptide-Based Vaccine in Participants With High-Risk Melanoma
Brief Title: Vaccine Therapy With or Without Imiquimod in Treating Patients Who Have Undergone Surgery for Stage II, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 11490; UVACC-MEL-45; UVACC-34204
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; sargramostim; Dimethyl Sulfoxide; Imiquimod; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: incomplete Freund's adjuvant
Biological: multi-epitope melanoma peptide vaccine
Biological: sargramostim
Biological: tetanus toxoid helper peptide
Drug: dimethyl sulfoxide
Drug: imiquimod
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Biological therapies, such as imiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. Giving vaccine therapy together with imiquimod after surgery may help the body kill any remaining tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects and best way to give vaccine therapy with or without imiquimod in treating patients who have undergone surgery for stage II, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of adjuvant transdermal vaccine therapy comprising multi-epitope melanoma peptides (MP), tetanus toxoid helper peptide (TET), and sargramostim (GM-CSF) in combination with Montanide ISA-51 or dimethyl sulfoxide with or without imiquimod in patients who have undergone surgical resection for stage II-IV melanoma.
* Determine, preliminarily, the immunogenicity of these regimens in these patients.
* Correlate, preliminarily, transdermal administration of these vaccines with the recruitment and maturation of epidermal Langerhans cells in these patients.
* Determine, preliminarily, the effects of timing of subsequent vaccine therapy comprising MP, TET, and GM-CSF emulsified in Montanide ISA-51, administered intradermally and subcutaneously, on the persistence of immune response in these patients.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive vaccine therapy comprising multi-epitope melanoma peptides (MP), tetanus toxoid helper peptide (TET), and sargramostim (GM-CSF) emulsified in Montanide ISA-51 transdermally (TD) on days 1, 8, and 15. Patients then receive the vaccine intradermally (ID) and subcutaneously (SC) on days 29, 50, 71, 92, 113, and 134.
* Arm II: Patients receive vaccine therapy as in arm I. Patients also receive imiquimod topically on days 0, 7, and 14.
* Arm III: Patients receive vaccine therapy comprising MP, TET, GM-CSF, and dimethyl sulfoxide TD on days 1, 8, and 15. Patients then receive vaccine therapy comprising MP, TET, and GM-CSF emulsified in Montanide ISA-51 ID and SC on days 29, 50, 71, 92, 113, and 134.
* Arm IV: Patients receive vaccine therapy as in arm III and imiquimod as in arm II.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3 and 5 weeks and then at disease progression.

PROJECTED ACCRUAL: A maximum of 26 patients (approximately 6 per treatment arm) will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed melanoma

  * Stage II-IV disease
* Has undergone surgical resection within the past 12 months

  * No clinical or radiological evidence of disease after surgical resection
  * Must have ≥ 1 undissected axillary and/or inguinal lymph node basin
* HLA-A1, -A2, or -A3 positive
* Ineligible for OR refused interferon

PATIENT CHARACTERISTICS:

Age

* 12 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Lactic dehydrogenase ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Hepatitis C negative

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Immunologic

* HIV negative
* No known or suspected allergy to any component of the study vaccines
* No autoimmune disorder with visceral involvement
* No prior active autoimmune disorder requiring cytotoxic or immunosuppressive therapy
* The following immunologic conditions are allowed:

  * Laboratory evidence of autoimmune disease (e.g., positive anti-nuclear antibody titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring non-steroidal anti-inflammatory drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 110 lbs
* No uncontrolled diabetes

  * Hemoglobin A1C < 7% (for patients with diabetes)
* No medical contraindication or potential problem that would preclude study compliance
* No known active addiction to alcohol or drugs
* No recent (within the past year) or ongoing illicit IV drug use

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior vaccinations that resulted in recurrent disease during or after vaccine administration allowed provided the last vaccination was administered more than 12 weeks ago
* Prior multi-epitope melanoma peptide vaccine that resulted in a negative immune response allowed
* More than 4 weeks since prior and no concurrent interferon (e.g., Intron-A®), interleukins (e.g., Proleukin®), or growth factors (e.g., Procrit®, Aranesp®, or Neulasta®)
* More than 4 weeks since prior and no concurrent allergy desensitization injections
* No influenza vaccine for at least 2 weeks before or after study vaccine administration

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas [e.g., carmustine or lomustine])
* No concurrent chemotherapy, including nitrosoureas

Endocrine therapy

* More than 4 weeks since prior and no concurrent oral or parenteral corticosteroids (e.g., prednisone)
* No prior or concurrent inhaled steroids (e.g., Advair®, Flovent®, Azmacort®)
* Concurrent topical corticosteroids allowed

Radiotherapy

* More than 4 weeks since prior and no concurrent radiotherapy
* Prior stereotactic radiosurgery allowed provided it was completed within the past 12 months

Surgery

* See Disease Characteristics
* More than 4 weeks since prior surgical resection of metastatic lesion(s)
* No concurrent surgery requiring general anesthesia

Other

* More than 4 weeks since prior and no other concurrent investigational agents
* More than 30 days since prior and no concurrent participation in another clinical study
* No other concurrent immunosuppressive therapy

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-11-04; Primary Completion 2006-07-28 (Actual); Study Completion 2006-07-28 (Actual)

PRIMARY OUTCOMES:
Safety if less than 33% of patients experience a dose-limiting at day 22

SECONDARY OUTCOMES:
Immune response by Elispot assay at day 22

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States